CLINICAL TRIAL: NCT00876655
Title: An Open-Label, Randomized, Single-Dose, 2-Treatment, 2-Sequence, Crossover, Exploratory Pharmacokinetic and Bioavailability Study of 2 Capsule Formulations of TR-701 (Torezolid Phosphate) in Normal Healthy Adults
Brief Title: Exploratory Pharmacokinetic and Bioavailability Study of 2 Capsule Formulations of Torezolid Phosphate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-025; TR701-108 (Other: TriusRX Unique ID)
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- free acid (Experimental): TR-701 free acid phosphate powder in capsule formulation (equivalent to 150 mg TR-700)
  Interventions: Drug: TR-701 free acid phosphate
- di-sodium phosphate salt (Experimental): One 200 mg capsule of TR-701 di-sodium phosphate salt (equivalent to 150 mg TR-700)
  Interventions: Drug: TR-701 di-sodium phosphate salt

INTERVENTIONS:
Drug: TR-701 di-sodium phosphate salt — One 200 mg capsule of TR-701 di-sodium phosphate salt (equivalent to 150 mg TR-700)
  Arms: di-sodium phosphate salt
Drug: TR-701 free acid phosphate — One 182 mg capsule of TR-701 free acid phosphate (equivalent to 150 mg TR-700)
  Arms: free acid

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of 2 different TR-701 oral formulations (free acid phosphate powder in capsule and di-sodium phosphate salt formulated capsule) after single doses in normal healthy adult subjects and to assess the relative bioavailability of TR-701 free acid phosphate powder in capsule formulation compared to di-sodium phosphate salt formulated capsule.

DETAILED DESCRIPTION:
Subjects will receive the following treatments in a crossover design:

Treatment A (Reference): One 200 mg capsule of TR-701 di-sodium phosphate salt (equivalent to 150 mg TR-700) administered orally after at least an 8-hour fast with 240 mL room temperature water;

Treatment B (Test): One 182 mg capsule of TR-701 free acid phosphate (equivalent to 150 mg TR-700) administered orally after at least an 8-hour fast with 240 mL room temperature water;

Descriptive statistics will be calculated for PK parameters including Cmax, Tmax, AUC0-t, and AUC0-inf.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs;
* Females will be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, surgically sterile for at least 90 days, or agree to use an acceptable form of contraception
* BMI of 18.5 to 32.0 kg/m2, inclusive

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* Pregnancy, lactation, or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics and relative bioavailability of TR-701 free acid phosphate powder in capsule formulation compared to di-sodium phosphate salt formulated capsule after single doses in normal healthy adult subjects | 4 days

SECONDARY OUTCOMES:
To determine the safety and tolerability of 2 different TR-701 oral formulations (free acid phosphate powder in capsule and di-sodium phosphate salt formulated capsule) after single doses in normal healthy adult | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: David C Carter, MD, Principal Investigator — Covance CRU
Locations (1):
- Covance Clinical Research Unit, Austin, Texas, United States

REFERENCES:
- [Derived] Flanagan SD, Bien PA, Munoz KA, Minassian SL, Prokocimer PG. Pharmacokinetics of tedizolid following oral administration: single and multiple dose, effect of food, and comparison of two solid forms of the prodrug. Pharmacotherapy. 2014 Mar;34(3):240-50. doi: 10.1002/phar.1337. Epub 2013 Aug 7. PMID 23926058